CLINICAL TRIAL: NCT05593354
Title: MicroPulse Transscleral Laser Therapy: A Prospective UK Study
Brief Title: MicroPulse TLT - UK Study
Acronym: MPTLTUKS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: IRIDEX Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21WE3716
Record Dates: First submitted 2022-10-17; First posted 2022-10-25 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Glaucoma; Glaucoma Eye; Glaucoma, Open-Angle; Glaucoma Secondary; Glaucoma, Angle-Closure; Glaucoma, Neovascular; Glaucoma Traumatic; Glaucoma Uveitic
Keywords: Glaucoma; Micropulse; Transscleral laser therapy; Cyclophotocoagulation
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Glaucoma, Neovascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- MPTLT patients: All UK patients undergoing MPTLT
  Interventions: Device: Micropulse Transscleral laser therapy

INTERVENTIONS:
Device: Micropulse Transscleral laser therapy — Transscleral laser cyclophotocoagulation using the IRIDEX Cyclo G6 machine
  Other Names: Cyclophotocoagulation; IRIDEX Cyclo G6

SUMMARY:
This Prospective Interventional Study will assess the efficacy of MPTLT in the UK.

DETAILED DESCRIPTION:
We are establishing a National Study of MPTLT procedures, co-ordinating with all UK treatment centres to capture prospectively, details of all MPTLT surgical procedure and outcomes. This will create a National UK Registry of MPTLT, allowing us to comply with NICE requirements while adding to the quality of evidence available to support this minimally invasive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma or ocular hypertension deemed clinically suitable for MPTLT treatment by their treating ophthalmologist; this includes but is not limited to (a) need for lower IOP, (b) need for fewer medications based on side effects, poor compliance, adverse effect on lifestyle or (c) evidence of disease progression based on function or structure
* Risk of invasive surgical procedure deemed too high by patient or surgeon
* Aged 18 years or older
* The ability to understand and comply with the trial consent process and procedures
* Willingness to be part of a national registry
* Ability to attend for follow-up
* Ability to give informed consent, or consent given by relative or carer

Exclusion Criteria:

* Clinical situations where in the opinion of the investigator, the ocular surface may be compromised by probe contact, including severe ocular surface inflammation
* Inability to give informed consent
* Unwillingness to have clinical data stored in a secure electronic format
* Inability to comply with the study or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UK patients with glaucoma or ocular hypertension deemed clinically suitable for MPTLT treatment by their treating ophthalmologist
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in intra-ocular pressure (IOP) following treatment | At the clinical visit closest to months 1, 3, 6, 12, 18, 24, 30 and 36
  Change in mean IOP before and after treatment, measured in mmHg using Goldmann Applanation Tonometry
Change in medication use following treatment | At the clinical visit closest to months 1, 3, 6, 12, 18, 24, 30 and 36
  Change in mean number of glaucoma medications before and after treatment

SECONDARY OUTCOMES:
Change in Retinal Nerve Fibre Layer (RNFL) following treatment | At the clinical visit closest to months 1, 3, 6, 12, 18, 24, 30 and 36
  RNFL thickness change, measured in micrometers using optical coherence tomography
Change in visual field (VF) following treatment | At the clinical visit closest to months 1, 3, 6, 12, 18, 24, 30 and 36
  Change in VF sensitivity, measured as mean deviation in dB units using computerised VF perimetry

OTHER OUTCOMES:
Compilation of evidence for further NICE review | 3 years
  To provide high quality evidence of treatment efficacy upon which to base a future review of the current NICE guidance, allowing subsequent treatments to be freely used in the UK, outside the context of research
Compliance with NICE recommendations | 3 years
  To allow continued use of MPTLT in the UK, whilst complying with NICE guidance, which currently recommends treatment only in the context of research

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Bloom, MB ChB FRCOphth, Principal Investigator — Imperial College Healthcare NHS Trust

IPD SHARING:
Plan to Share IPD: Undecided